CLINICAL TRIAL: NCT00888030
Title: P-cresol: Correlation With Glomerular Filtration Rate and Outcome in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, iwenwu, Attending physician, Chang Gung Memorial Hospital
Other Study IDs: IWW-0003
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Risk Factors; Renal Progression; Death
Keywords: p-cresol; indoxyl sulfate; chronic kidney disease; outcome
MeSH Terms: conditions — Death; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum level of p-cresol and indoxyl sulfate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 2: CKD patients with normal p-cresol
  Interventions: Other: there are no interventions currently listed for this study
- 3: CKD patient with normal indoxyl sulfate
  Interventions: Other: there are no interventions currently listed for this study
- 4: CKD patients with high indoxyl sulfate
  Interventions: Other: there are no interventions currently listed for this study
- 1: CKD patients with high p cresol
  Interventions: Other: there are no interventions currently listed for this study

INTERVENTIONS:
Other: there are no interventions currently listed for this study

SUMMARY:
End-stage renal disease is a global epidemia with an estimated incidence of 7% per year and high morbidity-mortality rate. Early detection of chronic kidney disease (CKD) and intervention for CKD complication is important to retard renal progression. However, "traditional uremic toxin" or "small water-soluble molecules" are poorly correlated with the renal function, uremic symptoms and outcomes of CKD patients.

Putative protein-bound solute, p-cresol, is accumulated in ESRD patients receiving dialysis therapy. This uremic solute was associated with endothelial dysfunction, immune dysregulation and can predict outcome in hemodialysis patient. P-cresol inhibits endothelial cell proliferation and endothelial response to inflammatory cytokines. In vitro, p-cresol decreases leukocyte transendotherliar migratory function and inhibit production of phagocyte reactive species. Clinically, p-cresol plays a pathophysiological role in the uremic toxicity. High free serum level of p-cresol is associated with mortality in hemodialysis patients.

Information of p-cresol in CKD patients is not available. The investigators hypothesized p-cresol can be accumulated in early CKD and have a positive correlation with the morbidity- mortality of CKD patients.

Value of p-cresol in different stages of CRF is still unknown. Information of p-cresol in CKD patients is not available. The investigators hypothesized p-cresol can be accumulated in early CKD and have a positive correlation with the morbidity- mortality of CKD patients.

The principal aim of this prospective cohort study is to investigate the association between total serum levels of p-cresol and the glomerular filtration rate. The correlation of level of p-cresol and morbidity-mortality in CKD patients will be also evaluated.

To determine the relationship, patients of nephrology clinic with a diagnosis of CKD were enrolled in this prospective study and follow-up for 1-year period. The association between total and free serum levels of p-cresol and the glomerular filtration rate were evaluated in CKD patients. The p-cresol level was correlated with other many inflammatory markers (white blood cell counts, ferritin, hs-crp, leptin) and also with the hospitalization rate secondary to cardiovascular and infectious event. The renal outcome and all-cause mortality was assessed. Determination of this relationship can help to establish an accurate marker for early detection of CKD and also its prognostic role in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* All CKD patients attended at out-patient department of nephrology were included for analysis.
* The inclusion criteria were adults aged > 18 y/o or < 80 y/o
* Estimated GFR or CCR < 60 ml/min
* No spontaneous renal improvement or progression in past 3 months.

Exclusion Criteria:

* Recent cardiovascular disease (Coronary artery disease, myocardial ischemia, cerebrovascular disease or peripheral artery disease) in past 3 months
* Recent infections requiring admission in past 3 months
* Uncontrolled hypertension
* Serum albumin level < 2.5mg/dL
* Unwilling to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All CKD patients attended at out-patient department of nephrology were included for analysis. The inclusion criteria were adults aged > 18 y/o or < 80 y/o; estimated GFR or CCR < 60 ml/min; no spontaneous renal improvement or progression in past 3 months.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
end stage renal disease, reduction of eGFR by 50% and death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iwen Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Nephrology,Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Background] Meijers BK, Bammens B, De Moor B, Verbeke K, Vanrenterghem Y, Evenepoel P. Free p-cresol is associated with cardiovascular disease in hemodialysis patients. Kidney Int. 2008 May;73(10):1174-80. doi: 10.1038/ki.2008.31. Epub 2008 Feb 27. PMID 18305466
- [Background] Atoh K, Itoh H, Haneda M. Serum indoxyl sulfate levels in patients with diabetic nephropathy: relation to renal function. Diabetes Res Clin Pract. 2009 Feb;83(2):220-6. doi: 10.1016/j.diabres.2008.09.053. Epub 2008 Nov 22. PMID 19027976
- [Background] Meijers BK, de Loor H, Verbeke K, Evenepoel P. p-Cresol for better or worse: but what are we measuring? Kidney Int. 2006 Jul;70(1):232; author reply 232-3. doi: 10.1038/sj.ki.5001530. No abstract available. PMID 16810293